CLINICAL TRIAL: NCT05906420
Title: Pc-ASTRAL Score for the Prediction of 3 Months Functional Outcome in Acute Ischemic Stroke at the Posterior Circulation
Brief Title: Posterior Circulation ASTRAL Prognostic Score
Status: Active, not recruiting | Type: Observational
Sponsor: University of Thessaly (Other)
Collaborators: University of Lausanne (Other); Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, George Ntaios, Professor of Internal Medicine George Ntaios, Aristotle University Of Thessaloniki
Other Study IDs: pc-ASTRAL
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Stroke Ischemic; Stroke Acute; Posterior Circulation Brain Infarction; Risk Score
MeSH Terms: conditions — Ischemic Stroke; Stroke; Brain Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (15):
- ASTRAL
  Interventions: Diagnostic Test: ASTRAL prognostic score
- Basel cohort
  Interventions: Diagnostic Test: ASTRAL prognostic score
- Berlin cohort
  Interventions: Diagnostic Test: ASTRAL prognostic score
- Bern Cohort
  Interventions: Diagnostic Test: ASTRAL prognostic score
- Bologna cohort
  Interventions: Diagnostic Test: ASTRAL prognostic score
- Dijon cohort
  Interventions: Diagnostic Test: ASTRAL prognostic score
- Lisbon cohort
  Interventions: Diagnostic Test: ASTRAL prognostic score
- Israel cohort
  Interventions: Diagnostic Test: ASTRAL prognostic score
- Innsbruck cohort
  Interventions: Diagnostic Test: ASTRAL prognostic score
- St. Gallen cohort
  Interventions: Diagnostic Test: ASTRAL prognostic score
- Lugano cohort
  Interventions: Diagnostic Test: ASTRAL prognostic score
- Chicago cohort
  Interventions: Diagnostic Test: ASTRAL prognostic score
- West Virginia cohort
  Interventions: Diagnostic Test: ASTRAL prognostic score
- Zurich cohort
  Interventions: Diagnostic Test: ASTRAL prognostic score
- Seoul cohort
  Interventions: Diagnostic Test: ASTRAL prognostic score

INTERVENTIONS:
Diagnostic Test: ASTRAL prognostic score — ASTRAL prognostic score

SUMMARY:
The goal of this study is to develop a prognostic score for ischemic posterior circulation strokes, based on our previous work on with the ASTRAL scores (Acute STroke Registry and Analysis of Lausanne) on overall stroke prognosis, intracranial occlusion, recanalization and stroke recurrences. The main question it aims to answer is the modified Rankin score in 3 months after the event.

Participants will be patients with acute ischemic stroke of the posterior circulation with mRS priot to event <3. All the data will be collected retrospectively from patients included in the ASTRAL registry between January 2003 and December 2021. The ASTRAL registry will be used as the derivation cohort of the score. Demographics, acute glucose, NIHSS score and acute imaging of each participant will be used from the derivation cohort in order to create an integer-based prognostic score. After internal validation, we plan to validate the score in external stroke registries to show its validity.

ELIGIBILITY:
Inclusion Criteria:

* Isolated posterior circulation strokes based on clinical or/and imaging evidence.
* Arriving within 24h at hospital since last proof of good health.

Exclusion Criteria:

* no available data for 3 months modified Rankin Score
* modified Rankin Score≥3 prior the event

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The participants included in this study are exclusively patients with acute ischemic stroke of the posterior circulation arriving at the hospital within 24h since last proof of good health. These patients must have a modified Rankin Score <3 prior the event and available data concerning: age, NIHSS, glucose levels at admission, mRS prior to event and 3 months after the event and acute phase imaging characteristics (CT and/or MRI) including large vessel occlusion, leukoaraiosis and ASPECTS score from the acute CT scan.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2003-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2025-11-24 (Estimated)

PRIMARY OUTCOMES:
3 months modified Ranking scale | January 2003-December 2021
  evaluation of 3 months neurological disability

CONTACTS AND LOCATIONS:
Locations (2):
- First Propedeutic Department of Internal Medicine & Stroke Unit, AHEPA University Hospital, Aristotle University of Thessaloniki, Thessaloniki, Central Macedonia, Greece
- Stroke Center, Department of clinical neurosciences, Lausanne University Hospital and University of Lausanne, Lausanne, Vaud Canton, Switzerland